CLINICAL TRIAL: NCT05360693
Title: Evaluation of Horizontal and Vertical Labial Bone Dimensional Changes After Flapless Immediate Implant Placement With and Without Bone Grafting: A 1-year Cone-beam Computed Tomography Randomized Clinical Trial.
Brief Title: Radiographic Evaluation of The Labial Bone Dimensional Changes After Immediate Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed Fouad Shemais, Lecturer in the department of Oral Medicine & Periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDCE.N1
Record Dates: First submitted 2022-04-30; First posted 2022-05-04 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Immediate Implants; Esthetic Zone; Labial Bone Dimensional Changes; Without Labial Bone Grafting; With Labial Grafting; Thin Labial Plate of Bone Pre-extraction
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant placement without bone grafting (Experimental): After atraumatic extraction of the non-restorable tooth using periotome and luxators, osteotomy site preparation will be done 3-5mm into the bone apical to the socket according to the manufacturer's instructions. Patients will receive an immediate post-extraction implant without any grafting material in the socket between the residual labial bone and implant surface.
  Interventions: Procedure: immediate implant placement without bone grafting
- immediate implant placement with bone grafting (Active Comparator): After atraumatic extraction of the non-restorable tooth using periotome and luxators, osteotomy site preparation will be done 3-5mm into the bone apical to the socket according to the manufacturer's instructions. Patients will receive an immediate post-extraction implant with placing bovine bone graft (Bio-oss) in the socket between the residual labial bone and implant surface.
  Interventions: Procedure: immediate implant placement with socket bone grafting

INTERVENTIONS:
Procedure: immediate implant placement without bone grafting — After atraumatic extraction of the non-restorable tooth using periotome and luxators, osteotomy site preparation will be done & patients will receive an immediate post-extraction implant without any grafting material in the socket between the residual labial bone and implant surface. After implant insertion, the labial bone dimensions of the buccal peri-implant defect will be measured using Automated Voxel Superimposition Method of CBCT scans. All the patients in this study had two scans; primary (preoperative) scan and secondary (Postoperative) scan, with standardization of the exposure parameters. All datafrom CBCT examinations were acquired in a DICOM format which were imported to OnDemand3D ®App software (Cybermed, Seoul, Korea). superimposition of DICOM sets of each patient using Fusion module of Ondemand 3D App software was done.
  Arms: immediate implant placement without bone grafting
Procedure: immediate implant placement with socket bone grafting — After atraumatic extraction of the non-restorable tooth using periotome and luxators, osteotomy site preparation will be done and patients will receive an immediate post-extraction implant with placing bovine bone graft (Bio-oss) in the socket between the residual labial bone and implant surface. After implant insertion, the labial bone dimensions of the buccal peri-implant defect will be measured using Automated Voxel Superimposition Method of CBCT scans. All the patients in this study had two scans; primary (preoperative) scan and secondary (Postoperative) scan, with standardization of the exposure parameters. All datafrom CBCT examinations were acquired in a DICOM format which were imported to OnDemand3D ®App software (Cybermed, Seoul, Korea). In order to ensure standardization and reproducibility of the CBCT cross sectional images used in this study, superimposition of DICOM sets of each patient using Fusion module of Ondemand 3D App software was done.
  Arms: immediate implant placement with bone grafting

SUMMARY:
For the dimension of the peri-implant buccal gap, a controversy is present whether complete bone formation labial to the implant. Therefore, leaving the blood clot in the large socket around implants without augmentation is questionable to result in complete bone fill and would not affect the buccal contour collapse. The aim of this clinical trial was to evaluate the labial bone dimensional changes after immediate implant placement in the esthetic zone with & without bone grafting inside the socket by using CBCT superimposition (Fusion) scans.

ELIGIBILITY:
inclusion criteria:

1. adult (>20 years) with non-restorable maxillary teeth in the esthetic zone,
2. thick gingival phenotype,
3. intact but thin labial plate of bone (≤1mm)
4. intact palatal bone extending at least 6mm apically,
5. sufficient apical bone to attain implant primary stability (a minimum of 35 Ncm insertion torque)
6. labio-palatal socket dimension measured from the CBCT axial cut at mid-crestal part ≥5mm.
7. patients agreed to sign a written informed consent.

Exclusion criteria:

1. smokers,
2. pregnant women,
3. patients with systemic disease,
4. patients with parafunctional habits such as bruxism or clenching,
5. infected socket,
6. periapical pathosis
7. history of radiotherapy or chemotherapy within the past 2 years.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Amount of bone labial to the implant | 1 year
  CBCT superimposition (fusion scans)
Horizontal labio-palatal bone width | 1 year
  CBCT superimposition (fusion scans)
horizontal labio-palatal bone collapse | 1 year
  CBCT superimposition (fusion scans)
vertical bone dimensional changes | 1 year
  CBCT superimposition (fusion scans)

SECONDARY OUTCOMES:
gingival index | 1 year
  bleeding on probing around customized healing abutments placed on the immediate implants
Implant failure | 1 year
  The following are the criteria of the implant success: the absence of mobility, the absence of acute or chronic peri-implant infection, the absence of radiolucency around the implant, without pocket probing depth (PPD) ≧ 5 mm, and without vertical bone loss ≧ 1.5 mm in the first year. The cases will be defined as failure if it can't reach any one of the success criteria.
Plaque Index | 1 year
  Plaque index
Postoperative Pain | 1 day, 3 days, 7 days
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: Noha A Ghallab, PhD, Principal Investigator — Professor of Oral Medicine & Periodontology; Ahmed I Abou- El-Fettouh, MSc, Study Director — Misr International University; Abdelrahman Zohny, BDs, Principal Investigator — Misr International University; Nael M Adel, BDs, Principal Investigator — Misr International University; Khaled Abdelghaffar, PhD, Study Chair — Professor of Periodontology, Ain Shams University; Mariam S Abdelmalak, BDs, Principal Investigator — Misr International University; Nesma M Shemais, PhD, Principal Investigator — Lecturer of Oral Medicine & Periodontology, Cairo University
Locations (2):
- Egypt (2):
  - International Dental Continuing Education, Cairo, Maadi
  - Faculty of Dentistry, Cairo University, Cairo, Manial

IPD SHARING:
Plan to Share IPD: No